CLINICAL TRIAL: NCT06214208
Title: Neuromodulation of Spinal Circuits: Effects on Spasticity, Nociception, and Motor Activation (Phase II)
Brief Title: Influence of Spinal Stimulation Frequency on Spasticity, Motor Control, and Pain After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Edelle Field-Fote, PT, PhD, Director, Spinal Injury Research & The Hulse Spinal Injury Laboratory, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2111327; 1R01HD101812-01A1 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30 Hz Frequency (Experimental): Intervention will be applied with a 30 Hz frequency.
  Interventions: Other: Transcutaneous Spinal Stimulation
- 50 Hz Frequency (Experimental): Intervention will be applied with a 50 Hz frequency.
  Interventions: Other: Transcutaneous Spinal Stimulation
- 80 Hz Frequency (Experimental): Intervention will be applied with an 80 Hz frequency.
  Interventions: Other: Transcutaneous Spinal Stimulation

INTERVENTIONS:
Other: Transcutaneous Spinal Stimulation — Transcutaneous spinal stimulation will be delivered for 30 minutes using biphasic pulses. A single cathode electrode will be placed over the skin of the back spine at the T11/T12 spinous interspace. Two reference electrodes will be placed over the stomach. Stimulation intensity will be set to 0.8x reflex threshold, as determined by posterior root muscle reflex testing before the intervention. Treatments will be a minimum of 72 hours apart.

SUMMARY:
The goal of this study is to identify the effect of different types of noninvasive spinal stimulation on spasticity (involuntary muscle activity), muscle strength, and pain in people with spinal cord injury. The spinal stimulation consists of electrical stimulation applied through one electrode over the skin of the lower back and two electrodes over the stomach. Testing will include participating in measurements before the intervention, during intervention, and immediately after the intervention. This study requires participants to come into Shepherd Center 4 consecutive days a week for 2-3 hours per day across 2-3 weeks.

DETAILED DESCRIPTION:
Transcutaneous spinal stimulation (TSS) is a noninvasive electrical stimulation that is applied over the skin of the low back and stomach. In prior research studies, TSS has reduced spasticity without the negative side effects of drug therapies. Although research in TSS is growing, the best dosage of TSS remains unknown. The investigators want to further advance the effects of TSS by comparing three different frequencies. Frequency is the number of electrical pulses that are delivered over a period of time. Frequency can affect the activation of nerves and therefore affect the outcome of TSS. Participation in this study includes testing of the participants' spasticity, strength, and pain before and after 30 minutes of TSS.

ELIGIBILITY:
Inclusion Criteria:

* Participants must agree to allow use of health information.
* Participants should be 16 years old or older.
* Participants must have had a spinal cord injury (SCI) of any severity (AIS A, B, C, or D) that happened at least 3 months ago.
* Objectively measurable spasticity in your legs.
* Participants must inform the investigators if there is a change in medications during the study.
* Participants must be able to follow instructions.
* Participants must be able to communicate if pain or discomfort is experienced.

Exclusion Criteria:

* People with spinal issues that are getting worse, such as degenerative or progressive vascular disorders.
* People neurological problems other than SCI.
* People with an injury level is below T12.
* People with un-treated or uncontrolled heart problems that the lead investigator believes could be affected by stimulation or affected by an increase in blood pressure.
* People with bone or joint problems that would make it hard to follow the study plan.
* Women who are pregnant or actively trying to become pregnant.
* People with implanted stimulators (like a baclofen pump, spinal stimulator, heart defibrillator, or diaphragmatic pacemaker)
* People with infection.
* People with skin that is broken or wounds in the area of the body where stimulation is applied.
* People who have or had certain types of cancer in the area of the body where stimulation will be applied.
* People who have had botulinum toxin or numbing shots in the test leg or spine in the last 6 months
* People who have had permanent spasticity treatment in the test leg or spine (like a certain type of surgery).
* Other health issues that the lead investigator things could make it unsafe for you to join the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Pendulum Test | 15 minutes
  During the pendulum test, the participant will be lying on a therapy mat with the lower leg hanging off the edge of the mat. A member of the study staff will support the participant's extended lower leg and then release the leg allowing it to swing freely. This test will be video recorded and the movement of the knee joint will be measured using software on the computer.

SECONDARY OUTCOMES:
Ankle Clonus Test | 15 minutes
  During the ankle clonus test, the participant will be seated at the edge of a mat with the lower leg hanging over the mat. A member of the study staff will support the participant's leg above a box and then release the leg allowing the front of the foot to land on the edge of the box. This test will be video recorded and the movement of the ankle joint will be measured using software on the computer.
Muscle activation | 20 minutes
  Participants will be asked to activate different leg muscles and produce the maximum amount of force possible. Muscle activation will be measured through sensors placed on the muscles and force production will be measured using a dynamometer.
Posterior root muscle reflexes | 25 minutes
  Posterior root muscle reflexes will be used to measure spinal reflex excitability. These reflexes will also be used to determine the intensity of stimulation that is applied during the intervention (0.8x soleus reflex threshold). During this test, participants have a single electrode over the skin of the back (T11/12) and two electrodes over the stomach (umbilicus). Brief pulses of stimulation will be applied at gradually increasing intensities while measuring muscle responses in different leg muscles.
Nociception/Pain | 15 minutes
  The investigators will measure nociception using the flexor reflex. The flexor reflex measures muscle responses to an unpleasant stimulus. Electrodes will be placed at the bottom of the foot. First, the investigators will measure muscle responses to a single stimulus (25 mA). Next, the investigators will measure muscle responses to 5 consecutive stimuli (25 mA). The investigators will then ask participants to rate the unpleasant stimulus on a scale of 0-10.
Quality of Spasticity Questionnaire | 5 minutes
  The Qualities of Spasticity Survey is a self-report questionnaire that asks participants about the physical qualities of their spasticity and how it impacts daily life. Participants will be asked to report experience with spasticity over the past 48 hours.
Modified Penn Spasm Frequency Scale | 2 minutes
  The Modified Penn Spasm Frequency Scale is a self-report questionnaire that asks participants to rate the frequency and severity of spasms during the last hour.
Stimulation Tolerability Questionnaire | 2 minutes
  Participants will be asked to rate how tolerable the spinal stimulation was during the session and to describe specific sensations that contributed to this rating.
Global Rating of Change Scale | 1 minute
  Participants will be asked to rate how much their change in spasticity affects their daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field-Fote, PT, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Inc., Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No